CLINICAL TRIAL: NCT07232472
Title: Wearable-enhanced Intervention for Elderly Depression and Sleep Disturbance - From Feasibility and Efficacy, to Development of the First Taiwanese Wearable-embedded Elderly Prospective Research Cohort
Brief Title: Wearable-Based Study of Depression and Sleep in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ta-wei Guu, Consultant Psychiatrist, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH114-REC2-068
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Elderly Depression; Sleep Disturbance
Keywords: wearable device; sleep disturbance; elderly depression; sleep; Photobiomodulation; Digital biomarkers
MeSH Terms: conditions — Parasomnias | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomised, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation (Experimental): Participants allocated to this arm will receive photobiomodulation for up to 8 weeks, using a wearable headband.
  Interventions: Device: Photobiomodulation
- sham (Sham Comparator): Participants allocated to this arm will not receive photobiomodulation for up to 8 weeks, using a sham wearable headband.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Photobiomodulation — A near-infrared photobiomodulation wearable device.
  Arms: Photobiomodulation
Device: Sham (No Treatment) — Participants allocated to this arm will receive neglectable photobiomodulation for up to 8 weeks, using a sham wearable headband.
  Arms: sham

SUMMARY:
This 4-year study aims to develop a safe and effective management model for late-life depression using wearable technologies. The research will recruit older adults (aged 60 and above) with major depressive disorder, confirmed by DSM-5 criteria.

In the first phase, participants will wear a research-grade actigraphy device (Geneactiv) for at least four weeks to assess its usability and accuracy compared with traditional questionnaires. In later phases, a double-blind randomized clinical trial will evaluate the efficacy of a photobiomodulation (PBM) headband in improving depressive and sleep symptoms.

The project will also establish Taiwan's first longitudinal database integrating wearable data, clinical symptoms, and biological markers, aiming to identify digital phenotypes and predictive biomarkers for elderly depression. The study is expected to advance precision psychiatry and digital health applications in geriatric mental health care.

DETAILED DESCRIPTION:
By 2025, Taiwan will become a super-aged society, with a rapidly growing number of older adults living with depression and related sleep problems. Late-life depression is often underdiagnosed and undertreated, and current assessments rely heavily on self-reported or clinician-rated questionnaires, which only provide snapshots of symptoms and may not accurately reflect daily variations in mood and sleep. These challenges highlight the urgent need for more objective, continuous, and accessible tools to monitor and manage depression in older adults.

Wearable devices, such as actigraphy and photobiomodulation (PBM), offer new opportunities for both assessment and intervention. Actigraphy can provide objective data on sleep-wake cycles, activity levels, and circadian rhythms, while PBM uses near-infrared light to modulate brain activity and improve mood and sleep quality. Building on our previous collaboration with Harvard University and recent findings from wearable PBM trials, this project seeks to establish an integrated, technology-assisted model for managing late-life depression in Taiwan.

This four-year project will begin by validating the feasibility and acceptability of a research-grade actigraphy device (Geneactiv) among older adults diagnosed with major depressive disorder (MDD). Objective activity and sleep data will be compared with questionnaire-based assessments to evaluate reliability and consistency, forming the foundation for Taiwan's first longitudinal wearable-based geriatric depression database.

In the second and third years, the study will conduct a double-blind, randomized, sham-controlled clinical trial to evaluate the safety and effectiveness of a wearable PBM headband device in improving depressive symptoms and sleep quality. Participants will continue their regular treatments while using the PBM device at home for daily sessions.

In the final year, longitudinal data from actigraphy, PBM intervention, clinical evaluations, and biological markers will be analyzed to identify digital phenotypes and predictive biomarkers associated with depression severity, treatment response, and functional outcomes. The long-term goal is to establish a comprehensive digital mental health platform that integrates biological, behavioral, and clinical dimensions, providing a scalable model for improving geriatric mental health in Taiwan's aging population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Major Depressive Disorder (MDD), either single or recurrent episode.
2. Have a Hamilton Depression Rating Scale (HAM-D, 17-item) total score of 14 or higher at baseline.
3. Participants who are currently taking medications that may affect mood, sleep, or circadian rhythms (e.g., antidepressants, sedative antipsychotics, or sleep aids) may be included, provided that the dosage has remained stable for at least two weeks prior to enrollment.
4. Prior to inclusion, informed consent must be obtained. If cognitive impairment prevents subjects from signing, consent may be obtained from their primary caregiver (who may be a legal or professional representative).

Exclusion Criteria:

1. Diagnosis of dementia of any severity, bipolar disorder, psychotic disorder, psychotic episode, or substance use disorder.
2. Active suicidal ideation or suicide attempt within the past three months.
3. Any other conditions deemed unsuitable for participation by the clinical physician, such as:

   * Currently experiencing acute delirium.
   * Suffering from respiratory infections, including COVID-19.
4. Participants with significant skin conditions on the head or conditions that could affect the efficacy of light therapy will be excluded. These include cases with:

   * Hemangiomas.
   * Scleroderma.
   * Psoriasis.
   * Rashes.
   * Open wounds.
   * Tattoos on the head. Additionally, individuals with head implants or those who have undergone photosensitizing drug treatments within two weeks prior to trial participation will also be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep and Circadian Rhythm | 8 weeks post-treatment.
  Sleep and circadian rhythm will be assessed using both questionnaire-based and device-based approaches.
  The questionnaire-based component will employ the Pittsburgh Sleep Quality Index (PSQI), which provides a total score ranging from 0 to 21, with lower scores indicating better sleep quality.
  The device-based component will analyze data from Geneactiv, processed with the validated open-source GGIR algorithm.
  1. Five sleep variables will be derived: sleep onset time, wake-up time, total sleep duration, sleep efficiency, and wake after sleep onset (WASO).
  2. Seven circadian rhythm variables will also be analyzed: light exposure amount and timing, M5/L5 (five-hour periods of highest/lowest activity), mean sleep midpoint time (MSA), intra-daily variability (IV), inter-daily stability (IS), daytime napping, and the Sleep Regularity Index (SRI).
Depression | 8 weeks post-treatment.
  Depression severity will be assessed using both questionnaire-based and device-based approaches. The questionnaire-based component will employ the depression severity assessed using the Hamilton Depression Rating Scale (HAM-D, 17-item version) which provides a total scores range from 0 to 52, with higher scores indicating more severe depressive symptoms. The device-based behavioral correlates (e.g., daytime activity, sleep fragmentation, light exposure regularity) derived from Geneactiv actigraphy will be analyzed to explore relationships with depressive symptom changes. Qualitative interviews will supplement quantitative findings to explore patient-reported mood changes and subjective well-being during the trial.
Feasibility, Acceptability, and User Experience of Device-Based Measurement and Management | From enrollment to the end of trial at 12 weeks
  Feasibility, satisfaction, and user experience with Geneactiv actigraphy and near-infrared photobiomodulation devices will be evaluated using:
  Quantitative assessments - Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST, Taiwanese version), compliance rate (measured by device-wearing duration and adherence), and completion rate of scheduled assessments.
  Qualitative interviews - conducted post-intervention to capture participants' experiences, perceived usability, and barriers to adoption.
  Data will be analyzed thematically to identify key factors affecting acceptability and implementation.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Beigang Hospital, London, Alabama, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We will decide if the IPD can be shared before the end of the study.

REFERENCES:
- [Result] Guu TW, Muurling M, Khan Z, Kalafatis C, Aarsland D, Ffytche D, Brem AK. Wearable devices: underrepresentation in the ageing society. Lancet Digit Health. 2023 Jun;5(6):e336-e337. doi: 10.1016/S2589-7500(23)00069-9. No abstract available. PMID 37236695
- [Result] Guu TW, Cassano P, Li WJ, Tseng YH, Ho WY, Lin YT, Lin SY, Chang JP, Mischoulon D, Su KP. Wearable, self-administered transcranial photobiomodulation for major depressive disorder and sleep: A randomized, double blind, sham-controlled trial. J Affect Disord. 2025 Mar 1;372:635-642. doi: 10.1016/j.jad.2024.12.065. Epub 2024 Dec 18. PMID 39706483